CLINICAL TRIAL: NCT01224171
Title: A Phase 3, Randomized, Placebo-Controlled, Blinded, Multicenter Study of the Induction of Clinical Response and Remission by Vedolizumab in Patients With Moderate to Severe Crohn's Disease
Brief Title: Study of Vedolizumab in Patients With Moderate to Severe Crohn's Disease
Acronym: GEMINI III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C13011; U1111-1158-2581 (Registry Identifier: WHO); 2009-016488-12 (EudraCT Number); NL34356.078.10 (Registry Identifier: CCMO)
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; LDP-02

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo intravenous infusion at Weeks 0, 2 and 6.
  Interventions: Other: Placebo
- Vedolizumab (Experimental): Participants received 300 mg intravenous vedolizumab at Weeks 0, 2, and 6.
  Interventions: Drug: vedolizumab

INTERVENTIONS:
Drug: vedolizumab — Vedolizumab for intravenous infusion
  Other Names: Entyvio; MLN0002; MLN02; LDP-02
  Arms: Vedolizumab
Other: Placebo — Placebo intravenous infusion
  Arms: Placebo

SUMMARY:
This study in patients with moderately to severely active Crohn's disease is designed to establish the efficacy and safety of vedolizumab for the induction of clinical response and remission.

DETAILED DESCRIPTION:
After completing the study, patients were eligible to enroll in a long term safety study with continued access to vedolizumab (study C13008; NCT00790933) if study drug was well tolerated, and no major surgical intervention for Crohn's disease occurred or was required.

Participants who did not enroll in Study C13008 were to complete the Final Safety visit (16 weeks after the last dose of study drug) for a maximum time on study of 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Diagnosis of moderately to severely active Crohn's disease
* Crohn's Disease involvement of the ileum and/or colon
* Demonstrated, over the previous 5 year period, an inadequate response to, loss of response to, or intolerance of at least one conventional therapy as defined by the protocol
* May be receiving a therapeutic dose of conventional therapies for inflammatory bowel disease (IBD) as defined by the protocol

Exclusion Criteria

* Evidence of abdominal abscess at the initial screening visit
* Extensive colonic resection, subtotal or total colectomy
* History of >3 small bowel resections or diagnosis of short bowel syndrome
* Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine
* Have received non permitted therapies within either 30 or 60 days, depending on the medication, as stated in the protocol
* Chronic hepatitis B or C infection; human immunodeficiency virus (HIV) infection
* Active or latent tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (41):
- United States (40):
  - Gastroenterology of the Rockies, Lafayette, Colorado
  - Gastroenterology Center of Connecticut P.C., Hamden, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Atlanta Gastroenterology Specialist PC, Suwanee, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Gastroenterology Associates, Baton Rouge, Louisiana
  - Gastroenterology Research of New Orleans, Hammond, Louisiana
  - Metropolitan Gastroenterology Group P.C., Chevy Chase, Maryland
  - Mid-Atlantic Medical Research Center, Hollywood, Maryland
  - Massachusetts General Hospital Crohn's and Colitis Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Minnesota Gastroenterology P.A., Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Long Island Clinical Research Associates, Great Neck, New York
  - New York Presbyterian Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology P.L.L.C, Charlotte, North Carolina
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - The Oregon Clinic-West Hills Gastroenterology, Portland, Oregon
  - Consultants in Gastroenterology, Columbia, South Carolina
  - Gastroenterology Center of the MidSouth PC, Germantown, Tennessee
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington School of Medicine, Seattle, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Zeidler Ledcor Center-Univerisity of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Sands BE, Van Assche G, Tudor D, Akhundova-Unadkat G, Curtis RI, Tan T. Vedolizumab in Combination With Corticosteroids for Induction Therapy in Crohn's Disease: A Post Hoc Analysis of GEMINI 2 and 3. Inflamm Bowel Dis. 2019 Jul 17;25(8):1375-1382. doi: 10.1093/ibd/izy384. PMID 30615117
- [Derived] Feagan BG, Sandborn WJ, Colombel JF, Byrne SO, Khalid JM, Kempf C, Geransar P, Bhayat F, Rubin DT. Incidence of Arthritis/Arthralgia in Inflammatory Bowel Disease with Long-term Vedolizumab Treatment: Post Hoc Analyses of the GEMINI Trials. J Crohns Colitis. 2019 Jan 1;13(1):50-57. doi: 10.1093/ecco-jcc/jjy125. PMID 30203005
- [Derived] Feagan BG, Lasch K, Lissoos T, Cao C, Wojtowicz AM, Khalid JM, Colombel JF. Rapid Response to Vedolizumab Therapy in Biologic-Naive Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2019 Jan;17(1):130-138.e7. doi: 10.1016/j.cgh.2018.05.026. Epub 2018 May 29. PMID 29857145
- [Derived] Colombel JF, Sands BE, Rutgeerts P, Sandborn W, Danese S, D'Haens G, Panaccione R, Loftus EV Jr, Sankoh S, Fox I, Parikh A, Milch C, Abhyankar B, Feagan BG. The safety of vedolizumab for ulcerative colitis and Crohn's disease. Gut. 2017 May;66(5):839-851. doi: 10.1136/gutjnl-2015-311079. Epub 2016 Feb 18. PMID 26893500
- [Derived] Rosario M, Dirks NL, Gastonguay MR, Fasanmade AA, Wyant T, Parikh A, Sandborn WJ, Feagan BG, Reinisch W, Fox I. Population pharmacokinetics-pharmacodynamics of vedolizumab in patients with ulcerative colitis and Crohn's disease. Aliment Pharmacol Ther. 2015 Jul;42(2):188-202. doi: 10.1111/apt.13243. Epub 2015 May 20. PMID 25996351
- [Derived] Sands BE, Feagan BG, Rutgeerts P, Colombel JF, Sandborn WJ, Sy R, D'Haens G, Ben-Horin S, Xu J, Rosario M, Fox I, Parikh A, Milch C, Hanauer S. Effects of vedolizumab induction therapy for patients with Crohn's disease in whom tumor necrosis factor antagonist treatment failed. Gastroenterology. 2014 Sep;147(3):618-627.e3. doi: 10.1053/j.gastro.2014.05.008. Epub 2014 May 21. PMID 24859203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately to severely active Crohn's Disease took part in the study at 107 sites worldwide from 24 November 2010 to 12 April 2012. Approximately 75% of participants were to have previously failed tumor necrosis factor alpha (TNFα) antagonist therapy and approximately 25% were to have been naïve to TNFα antagonist therapy.
Pre-assignment Details: Participants were randomized 1:1 to receive either 300 mg vedolizumab or placebo. Randomization to treatment assignment was stratified by the presence or absence of previous failure of TNFα antagonist therapy or naïve to TNFα antagonist therapy, concomitant use of oral corticosteroids and concomitant use of immunomodulators.
Period: Overall Study
Arm/Group | Placebo | Vedolizumab
Started | 207 | 209
TNFα Antagonist Failure Population | 157 (Previously failed (inadequate response, loss of response, or intolerance) TNFα antagonist therapy) | 158 (Previously failed (inadequate response, loss of response, or intolerance) TNFα antagonist therapy)
Completed | 192 (Completed study is defined as patients who completed the Week 10 assessments.) | 196 (Completed study is defined as patients who completed the Week 10 assessments.)
Not Completed | 15 | 13
Not completed — Adverse Event | 8 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 5 | 1
Not completed — Withdrawal of Consent | 2 | 4
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Overall Intent-to-treat (ITT) Population consisted of all randomized participants who received any amount of blinded study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vedolizumab | Total
Number analyzed (Participants) | 207 | 209 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (13.15) | 38.6 (12.14) | 37.9 (12.66)
Age, Customized [Number; unit: participants]
  < 35 years | 105 | 88 | 193
  ≥ 35 years | 102 | 121 | 223
Age, Customized [Number; unit: participants]
  < 65 years | 202 | 206 | 408
  ≥ 65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 118 | 236
  Male | 89 | 91 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 199 | 204 | 403
  Unknown or Not Reported | 4 | 1 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 186 | 188 | 374
  Black | 5 | 4 | 9
  Asian | 9 | 9 | 18
  Other | 7 | 6 | 13
  Not Reported | 0 | 2 | 2
Body Weight [Mean (Standard Deviation); unit: kg] | 71.3 (19.22) | 69.5 (17.76) | 70.4 (18.50)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (6.13) | 24.0 (5.13) | 24.3 (5.65)
Geographic Region [Number; unit: participants]
  North America | 95 | 102 | 197
  Western/Northern Europe | 37 | 38 | 75
  Central Europe | 46 | 41 | 87
  Eastern Europe | 15 | 10 | 25
  Asia/Australia/Africa | 14 | 18 | 32
Duration of Crohn's Disease (CD) [Mean (Standard Deviation); unit: years] | 10.0 (7.98) | 10.6 (8.75) | 10.3 (8.37)
Duration of Crohn's Disease - Categorical [Number; unit: participants]
  < 1 year | 12 | 11 | 23
  ≥ 1 to < 3 years | 25 | 28 | 53
  ≥ 3 to < 7 years | 52 | 52 | 104
  ≥ 7 years | 118 | 118 | 236
Baseline Disease Activity - Crohn's Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: units on a scale] — Baseline disease activity represents the baseline CDAI score. The CDAI is a numerical calculation derived from the sum of products from a list of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to ~600 points with lower scores indicating disease remission and higher scores indicating disease worsening.
  units on a scale | 301.3 (54.97) | 313.9 (53.17) | 307.7 (54.38)
Baseline Disease Activity - Categorical [Number; unit: participants]
  CDAI ≤ 330 | 148 | 132 | 280
  CDAI > 330 | 59 | 77 | 136
C-reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] | 18.5 (21.98) | 19.0 (23.17) | 18.8 (22.56)
CRP - Categorical [Number; unit: participants]
  ≤ 2.87 mg/L | 41 | 46 | 87
  > 2.87 to ≤ 5 mg/L | 19 | 14 | 33
  > 5 to ≤ 10 mg/L | 42 | 48 | 90
  > 10 mg/L | 105 | 101 | 206
Fecal Calprotectin [Mean (Standard Deviation); unit: μg/g] — Number of participants for whom baseline fecal calprotectin data were available were 206 and 204, respectively.
  μg/g | 1426.5 (2357.76) | 1148.1 (1878.58) | 1288.0 (2134.79)
Fecal Calprotectin - Categorical [Number; unit: participants]
  ≤ 250 μg/g | 47 | 52 | 99
  > 250 to ≤ 500 μg/g | 35 | 35 | 70
  > 500 μg/g | 124 | 117 | 241
  Missing | 1 | 5 | 6
Disease Localization [Number; unit: participants]
  Ileum only | 29 | 33 | 62
  Colon only | 52 | 48 | 100
  Ileocolonic (both ileum and colon) | 126 | 128 | 254
History of Prior Surgery for Crohn's Disease [Number; unit: participants]
  Yes | 89 | 92 | 181
  No | 118 | 117 | 235
Smoking Status [Number; unit: participants]
  Current Smoker | 58 | 65 | 123
  Never Smoked | 102 | 93 | 195
  Former Smoker | 47 | 51 | 98
History of Fistulizing Disease [Number; unit: participants]
  Yes | 77 | 71 | 148
  No | 130 | 138 | 268
Draining Fistula at Baseline [Number; unit: participants]
  Yes | 25 | 25 | 50
  All Closed | 0 | 1 | 1
  No Fistula | 182 | 183 | 365
Extraintestinal Manifestations at Baseline [Number; unit: participants]
  Yes | 130 | 116 | 246
  No | 77 | 93 | 170

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Remission in the Tumor Necrosis Factor Alpha (TNFα) Antagonist Failure Subpopulation
Description: Clinical remission is defined as a Crohn's Disease Activity Index (CDAI) score ≤ 150 points.
  The CDAI is used to quantify the symptoms of patients with Crohn's disease and consists of eight factors, each summed after adjustment with a weighting factor. The components of the CDAI are:
  * Number of liquid or soft stools each day for 7 days;
  * Abdominal pain (graded from 0-3 on severity) each day for 7 days;
  * General well-being, subjectively assessed from 0 (well) to 4 (terrible) each day for 7 days;
  * Presence of complications;
  * Taking Lomotil or opiates for diarrhea;
  * Presence of an abdominal mass (0 as none, 2 as questionable, 5 as definite);
  * Hematocrit of < 0.47 in men and < 0.42 in women;
  * Percentage deviation from standard weight.
  The total score ranges from 0 to approximately 600 and with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving clinical remission.
Time Frame: Week 6
Population: TNFα Antagonist Failure Intent-to-treat (ITT) subpopulation which consisted of all randomized participants who received any amount of blinded study drug who met the TNFα antagonist failure criterion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab
Number analyzed (Participants) | 157 | 158
percentage of participants | 12.1 [7.0 to 17.2] | 15.2 [9.6 to 20.8]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab; Clinical remission was tested using the Cochran-Mantel-Haenszel (CMH) chi-square test at a 5% significance level with stratification according to concomitant use of oral corticosteroids and concomitant use of immunomodulators (6-mercaptopurine [6-MP], azathioprine, or methotrexate) for the TNFα antagonist failure subpopulation; Test type: Superiority or Other; p = 0.4332, Cochran-Mantel-Haenszel; Risk Difference (RD) = 3.0, 95% CI 2-sided [-4.5 to 10.5] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo

2. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 6 in the Overall Population
Description: as for outcome 1
Time Frame: Week 6
Population: Overall ITT population, consisting of all randomized participants who received any amount of blinded study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab
Number analyzed (Participants) | 207 | 209
percentage of participants | 12.1 [7.6 to 16.5] | 19.1 [13.8 to 24.5]

3. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 10 in the TNFα Antagonist Failure Subpopulation
Description: as for outcome 1
Time Frame: Week 10
Population: TNFα Antagonist Failure Intent-to-treat (ITT) Subpopulation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab
Number analyzed (Participants) | 157 | 158
percentage of participants | 12.1 [7.0 to 17.2] | 26.6 [19.7 to 33.5]

4. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 10 in the Overall Population
Description: as for outcome 1
Time Frame: Week 10
Population: Overall ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab
Number analyzed (Participants) | 207 | 209
percentage of participants | 13.0 [8.5 to 17.6] | 28.7 [22.6 to 34.8]

5. Secondary Outcome: Percentage of Participants With Sustained Clinical Remission in the TNFα Antagonist Failure Population
Description: Sustained clinical remission is defined as a CDAI score ≤ 150 points at both Week 6 and Week 10. The CDAI is used to quantify the symptoms of patients with Crohn's disease and consists of eight factors, each summed after adjustment with a weighting factor. The components of the CDAI are:
  * Number of liquid or soft stools each day for 7 days;
  * Abdominal pain (graded from 0-3 on severity) each day for 7 days;
  * General well-being, subjectively assessed from 0 (well) to 4 (terrible) each day for 7 days;
  * Presence of complications;
  * Taking Lomotil or opiates for diarrhea;
  * Presence of an abdominal mass (0 as none, 2 as questionable, 5 as definite);
  * Hematocrit of < 0.47 in men and < 0.42 in women;
  * Percentage deviation from standard weight.
  The total score ranges from 0 to approximately 600 and with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving sustained clinical remission.
Time Frame: Week 6 and Week 10
Population: TNFα Antagonist Failure ITT Subpopulation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab
Number analyzed (Participants) | 157 | 158
percentage of participants | 8.3 [4.0 to 12.6] | 12.0 [7.0 to 17.1]

6. Secondary Outcome: Percentage of Participants With Sustained Clinical Remission in the Overall Population
Description: as for outcome 5
Time Frame: Week 6 and Week 10
Population: Overall ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab
Number analyzed (Participants) | 207 | 209
percentage of participants | 8.2 [4.5 to 12.0] | 15.3 [10.4 to 20.2]

7. Secondary Outcome: Percentage of Participants With Enhanced Clinical Response at Week 6 in the TNFα Antagonist Failure Subpopulation
Description: Enhanced clinical response is defined as a ≥ 100-point decrease in CDAI score from Baseline.
  The CDAI is used to quantify the symptoms of patients with Crohn's disease and consists of eight factors, each summed after adjustment with a weighting factor. The components of the CDAI are:
  * Number of liquid or soft stools each day for 7 days;
  * Abdominal pain (graded from 0-3 on severity) each day for 7 days;
  * General well-being, subjectively assessed from 0 (well) to 4 (terrible) each day for 7 days;
  * Presence of complications;
  * Taking Lomotil or opiates for diarrhea;
  * Presence of an abdominal mass (0 as none, 2 as questionable, 5 as definite);
  * Hematocrit of < 0.47 in men and < 0.42 in women;
  * Percent deviation from standard weight.
  The total score ranges from 0 to approximately 600 and with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving enhanced clinical response.
Time Frame: Baseline and Week 6
Population: TNFα Antagonist Failure ITT Subpopulation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab
Number analyzed (Participants) | 157 | 158
percentage of participants | 22.3 [15.8 to 28.8] | 39.2 [31.6 to 46.9]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a patient administered a pharmaceutical product, which did not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) was any AE, occurring at any dose and regardless of causality that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was an important medical event based upon appropriate medical judgment that may have jeopardized the patient and may have required medical or surgical intervention to prevent 1 of the outcomes listed above, or any diagnosis of progressive multifocal leukoencephalopathy (PML).
  Relationship to study drug administration was determined by the investigator responding yes or no to the question: Is there a reasonable possibility that the AE is associated with the study drug?
Time Frame: From the date of first study drug administration to Week 22, through the 14 March 2012 database lock date. At the time of this database lock, 7 patients had completed Week 10 or early termination assessments but not Week 22 assessments.
Population: Overall Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Vedolizumab
Number analyzed (Participants) | 207 | 209
participants
  Any adverse event | 124 | 117
  Drug-related adverse event | 34 | 34
  Adverse event resulting in study discontinuation | 8 | 4
  Serious adverse event | 16 | 13
  Serious infection adverse event | 0 | 2
  Drug-related serious adverse event | 1 | 1
  Serious adverse event resulting in discontinuation | 5 | 4
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of first study drug administration to Week 22, through the 14 March 2012 database lock date. At the time of this database lock, 7 patients had completed Week 10 or early termination assessments but not Week 22 assessments.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vedolizumab
Serious Adverse Events (participants affected / at risk) | 16/207 | 13/209
Other Adverse Events (participants affected / at risk) | 29/207 | 25/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=207) | Vedolizumab (N=209)
Crohn's disease (Gastrointestinal disorders) | 11 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Demyelination (Nervous system disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=207) | Vedolizumab (N=209)
Nausea (Gastrointestinal disorders) | 5 | 12
Headache (Nervous system disorders) | 15 | 11
Pyrexia (General disorders) | 13 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.